CLINICAL TRIAL: NCT06007352
Title: Use of Antibiotic Based Irrigation for Ureteroscopic Treatment of Urolithiasis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding issue
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000035721; 000 (Other: CTGTY)
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Urinary Tract Infections; Sepsis
Keywords: UTI; Gentamicin; Ureteroscopy
MeSH Terms: conditions — Urinary Tract Infections; Sepsis | interventions — Gentamicins

STUDY DESIGN:
Intervention Model Description: phase II, parallel randomized control trial with 1:1 allocation
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Gentamicin-Based Irrigation (Experimental): This group will receive 120 mg of Gentamicin in 3 L NaCl as irrigation fluid during ureteroscopy
  Interventions: Drug: Gentamicin
- 3 L NaCl Irrigation (Placebo Comparator): This group will receive the typical NaCl irrigation used during ureteroscopy
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Gentamicin — Participants will be given 120 mg of gentamicin infused in 3 L NaCl used in irrigation for ureteroscopy
  Arms: Gentamicin-Based Irrigation
Other: Placebo — 3 L of NaCl irrigation typically used for ureteroscopy surgery
  Arms: 3 L NaCl Irrigation

SUMMARY:
The purpose of the study is to investigate whether the use of gentamicin-based irrigation fluid during ureteroscopy decreases the risk of UTIs and other post-operative infections after surgery.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether the utilization of gentamicin-based irrigation fluid during ureteroscopy decreases the rate of 30-day post-operative symptomatic urinary tract infections in patients at higher risk of urinary tract infection undergoing stone surgery for urolithiasis.

The secondary objectives of this study are to determine whether the utilization of gentamicin-based irrigation fluid during ureteroscopy affects the 30-day post-operative rates of patient-initiated telephone calls, readmission rates, urosepsis rates based on SIRS criteria, and overall post-operative oral/intravenous antibiotic administration.

In this prospective study, 120 mg of gentamicin prepared in 3 liters of normal saline will be used as irrigation during ureteroscopic surgery for urolithiasis. At this concentration, 40 μg/mL, the MBC would be achieved for pathogenic urogenital bacteria. Due to the concerns of nephrotoxicity and ototoxicity at higher doses of gentamicin, in the unlikely event of complete pyelo-venous backflow, the intravenous circulation of 120 mg of gentamicin would be less than the surgical prophylaxis intravenous dosing for patients weighing more than 60 kg. For the single intravenous dose for surgical prophylaxis, post-operative monitoring of renal function, and gentamicin peak and trough levels are not routinely obtained.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Diagnosed with urolithiasis (obstructing ureteral stone, large non-obstructing renal stones) warranting surgical intervention in line with American Urological Association guidelines for urolithiasis
* At a higher risk for infectious complications following ureteroscopy based on a history of atleast one of the below:
* 3 more urinary tract infections over 12 month period not on suppressive antibiotic therapy
* Prior infectious complication following ureteroscopy
* Placement of ureteral stent in the setting of obstructing ureteral stone with concern for superimposed urinary tract infection
* Positive pre-operative urine culture treated with culture-appropriate antimicrobial therapy
* Planned for cystoscopy, ureteroscopy with possible laser lithotripsy, and ureteral stent placement
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 8 weeks after the end of gentamicin administration. Female patients of reproductive potential will have pregnancy screen prior to surgery per standard operating room protocol.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner

Exclusion Criteria:

* Estimated Glomerular Filtration Rate less than 60 mL/min
* History of sensorineural hearing loss, vertigo, idiopathic dizziness
* Active pregnancy or currently lactating
* Known allergic reactions to components of gentamicin
* Administration of intravenous gentamicin as part of surgical antibiotic prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Symptomatic urinary tract infection | Within 30 days of surgery
  Development of a symptomatic urinary tract infection after surgery

SECONDARY OUTCOMES:
Urosepsis | Within 30 days of surgery
  Development of urosepsis after URS based on SIRS criteria
Re-admission to hospital | Within 30 days of surgery
  Re-admission to hospital after surgery for any reason
Patient self-reported symptoms | within 30 days of surgery
  Self-reported symptoms after the operation of the following: new hearing loss, vertigo and dizziness

CONTACTS AND LOCATIONS:
Overall Officials: Piruz Motamedinia, M.D., Principal Investigator — Yale School of Medicine, Department of Urology
Locations (1):
- Yale New Haven Health, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No